CLINICAL TRIAL: NCT03443219
Title: A Prospective Randomised Controlled Trial of the LMA Supreme™ Versus the Spritztube® Tracheal Cannula in Anesthetized Adult Patients
Brief Title: RCT- LMA Supreme™ Versus the Spritztube® Tracheal Cannula in Anesthetized Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Principal Investigator, Silvia De Rosa, Medical Doctor, St. Bortolo Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 29/16
Record Dates: First submitted 2018-02-12; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Airway Management
Keywords: Airway Management; Extraglottic airway device; Laryngeal mask airway; Spritztube

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: opening a sealed envelope, provided by an independent physician blinded to patient's allocation In addition, outcome assessor were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spritztube® (Experimental): The patients were randomly allocated to two groups by using computer-generated numbers.In Spritztube® group, Spritztube® was inserted into each patient after anesthesia induction.
  Interventions: Device: Spritztube®
- LMA Supreme™ (Active Comparator): The patients were randomly allocated to two groups by using computer-generated numbers.In vgroup, LMA Supreme™was inserted into each patient after anesthesia induction.
  Interventions: Device: LMA Supreme™

INTERVENTIONS:
Device: Spritztube® — After preoxygenation, anaesthesia was induced with midazolam, propofol, and fentanyl,Spritztube® was inserted and both cuffs inflated
  Arms: Spritztube®
Device: LMA Supreme™ — After preoxygenation, anaesthesia was induced with midazolam, propofol, and fentanyl,LMA Supreme™ was inserted and both cuffs inflated
  Arms: LMA Supreme™

SUMMARY:
The study compares the LMA Supreme™ versus the Spritztube® tracheal cannula in anesthetized adult patients.

The current randomized study is designed to assess the success placement of blind insertion using LMA Supreme™ , in comparison with the Spritztube® tracheal cannula.

In addition, time, number of attempts, easy insertion and the number of complications at insertion and removal will be assessed.

The investigators hypothesize that the LMA Supreme™ versus the Spritztube® tracheal cannula will similarly perform during anesthetized adult patients despite differences in their structural design.

DETAILED DESCRIPTION:
A new extraglottic airway device, the Spritztube® [tracheal cannula, Med Europe s.r.l], was developed combining the ability to perform both EAD ventilation and oro-tracheal fibreoptic intubation using the same device. The Spritztube® consists of a silicone cannula with two low-pressure cuffs: a proximal cuff, designed to seal the pharynx cranially of the epiglottis and a distal cuff, designed to seal the oesophagus. The positioning of this device requires the aid of a spindle, that keep the cuffs on the same line and it is rigid enough to allow the passage through oropharynx tissue. That can be inserted blindly as extraglottic device or through the use of direct laryngoscopy or fibroscopy as tracheal cannula.

The current randomized study is designed to assess the success placement of blind insertion using LMA Supreme™ , in comparison with the Spritztube® tracheal cannula.

In addition, time, number of attempts, easy insertion and the number of complications at insertion and removal will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status classification I, II, and III;
* Age > 18 years
* Elective surgery in the supine position

Exclusion Criteria:

* Pregnancy
* Age <18 years
* Not eligibility for surgery
* Predicted difficult airway management
* Positive history for esophageal or pharyngeal diseases
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
the successful placement of device in two groups | Intraoperative
  A successful intubation attempt was recognized if the breathing circuit was connected, the breath sounds over the lung were present and the End tidal CO2 trace was revealed.

SECONDARY OUTCOMES:
Insertion time (in seconds) | Intraoperative
  The insertion time was measured from the insertion of device into the patient's mouth to connecting the breathing circuit.
Number of attempts | Intraoperative
  If placement had failed after three attempts, the study was abandoned and the airway was maintained through a tracheal tube.
Easy to insert | Intraoperative
  A successful insertion of device in just one attempt
number of complications at insertion | Intraoperative
  air leak at induction, laryngospasm, obstruction after induction, gastric insufflation, failure device
number of complications at removal | Postoperative
  dysphagia, hoarseness and sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Bonato, MD, Study Director — Department of Anesthesiology and Intensive Care, San Bortolo Hospital, Vicenza, Italy

REFERENCES:
- [Derived] De Rosa S, Messina A, Sorbello M, Rigobello A, Colombo D, Piccolo A, Bonaldi E, Gennaro P, Urukalo V, Pellizzari A, Bonato R, Carboni SC. Laryngeal Mask Airway Supreme vs. the Spritztube tracheal cannula in anaesthetised adult patients: A randomised controlled trial. Eur J Anaesthesiol. 2019 Dec;36(12):955-962. doi: 10.1097/EJA.0000000000001106. PMID 31644512